CLINICAL TRIAL: NCT02950220
Title: A Phase I/Ib Study of the PD-1 Antibody Pembrolizumab in Combination With Ibrutinib in Relapsed/Refractory Non-Hodgkin's Lymphoma (NHL)
Brief Title: Pembrolizumab and Ibrutinib in Treating Patients With Relapsed or Refractory Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kami Maddocks (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Kami Maddocks, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-16070; NCI-2016-01560 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA016058 (NIH)
Record Dates: First submitted 2016-10-28; First posted 2016-11-01 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: B-Cell Lymphoma, Unclassifiable, With Features Intermediate Between Diffuse Large B-Cell Lymphoma and Classical Hodgkin Lymphoma; Grade 1 Follicular Lymphoma; Grade 2 Follicular Lymphoma; Grade 3a Follicular Lymphoma; Mediastinal Lymphoma; Recurrent B-Cell Non-Hodgkin Lymphoma; Recurrent Burkitt Lymphoma; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Follicular Lymphoma; Recurrent Lymphoplasmacytic Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Waldenstrom Macroglobulinemia; Refractory B-Cell Non-Hodgkin Lymphoma; Refractory Burkitt Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory Follicular Lymphoma; Refractory Lymphoplasmacytic Lymphoma; Refractory Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Follicular; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell; Waldenstrom Macroglobulinemia | interventions — ibrutinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Ibrutinib; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase I/Ib trial studies the side effects and best dose of ibrutinib when given together with pembrolizumab and to see how well they work in treating patients with non-Hodgkin lymphoma that has come back or does not respond to treatment. Monoclonal antibodies, such as pembrolizumab, may interfere with the ability of cancer cells to grow and spread. Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Given pembrolizumab and ibrutinib may work better in treating patients with non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of the combination of ibrutinib and pembrolizumab in patients with relapsed/refractory non-Hodgkin lymphoma (NHL).

II. To determine the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) of the combination of ibrutinib and pembrolizumab in patients with relapsed/refractory NHL.

III. To evaluate the efficacy of the combination of ibrutinib and pembrolizumab in patients with relapsed/refractory NHL.

SECONDARY OBJECTIVES:

I. To determine the overall response rate (ORR), duration of response, progression-free survival and overall survival of the combination of ibrutinib and pembrolizumab in patients with relapsed/refractory NHL.

TERTIARY OBJECTIVES:

I. To explore the relationship between prognostic parameters including ki-67 staining, PD-1 staining and cell of origin (activated B-cell or ABC versus germinal center B-cell or GCB) with ORR to the combination of ibrutinib and pembrolizumab in patients with relapsed/refractory NHL.

II. To determine relationship between gene mutations and resistance to therapy with the combination of ibrutinib and pembrolizumab in patients with relapsed/refractory NHL (BTK, PLC gamma 2, PD-1).

III. To evaluate and monitor effects on B-, T-, and natural killer (NK)-cell function with the combination of ibrutinib and pembrolizumab in patients with relapsed/refractory NHL.

OUTLINE: This is a phase I, dose-escalation study of ibrutinib followed by a phase Ib study.

Patients receive ibrutinib orally (PO) daily on days 1-21 and pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 21 days for up to 17 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days, and then every 3 months for 2 years and every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed B-cell NHL with any of the following subtypes: diffuse large B-cell lymphoma (DLBCL), mantle cell lymphoma (MCL), follicular lymphoma (FL), marginal zone lymphoma (MZL) and lymphoplasmacytic lymphoma/Waldenstrom's macroglobulinemia (LL/WM), Burkitt's lymphoma (BL); patients with histological transformation to DLBCL from indolent lymphoma, primary mediastinal lymphoma and grey zone lymphoma are eligible (Part 1)
* Patients must have received at least one prior therapy; prior autologous stem cell transplant is permitted; patients with DLBCL who have not had prior high-dose therapy (HDT)/autologous stem cell transplant (ASCT) must be ineligible for transplant; prior ibrutinib is not permitted if patients have progressed on therapy (Part 1)
* Patients with Waldenstrom's macroglobulinemia (WM) must meet the indications for treatment per the International Workshop on Waldenstrom's Macroglobulinemia (IWWM) (Part 1)
* Histologically confirmed B-cell NHL (Part 2):

  * Group 1: with only de novo DLBCL,
  * Group 2: with only FL of grade 1, 2 or 3a
  * Group 3: with only MCL with t(11;14) or overexpression of cyclin D1
  * Group 4: all other NHL including MZL, LL, WM, BL, primary mediastinal B cell lymphoma (PMBCL), gray zone lymphoma (GZL) and patients with histological transformation to DLBCL from indolent lymphoma are eligible
* Patients must have received at least one prior therapy; prior autologous stem cell transplant is permitted; patients with DLBCL who have not had prior HDT/ASCT must be ineligible for transplant; prior ibrutinib is not permitted if patients have progressed on therapy (Part 2)
* Patients with Waldenstrom's macroglobulinemia (WM) must meet the indications for treatment per the International Workshop on Waldenstrom's Macroglobulinemia (IWWM) (Part 2)
* Be willing and able to provide written informed consent/assent for the trial
* Have evaluable disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Absolute neutrophil count (ANC) >= 1,000/mcL
* Platelets >= 50,000/mcL in the absence of transfusion support within 7 days of determining eligibility
* Hemoglobin >= 8 g/dL
* Serum creatinine =< 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) OR >= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN
* Serum total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN
* Aspartate aminotransferases (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X ULN OR =< 5 X ULN for subjects with liver metastases
* Albumin >= 2.5 mg/dL
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment; subjects may use topical or inhaled corticosteroids or low-dose steroids (=< 10 mg of prednisone or equivalent per day) as therapy for comorbid conditions; during study participation, subjects may receive systemic or enteric corticosteroids as needed for treatment-emergent comorbid conditions
* Has a known history of active TB (Bacillus tuberculosis)
* Hypersensitivity to pembrolizumab or ibrutinib or any of their excipients
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has had prior chemotherapy or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent

  * Note: subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
  * Note: if subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy; patients must be 4 weeks out from major procedures and 2 weeks out from minor procedures
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has known active central nervous system (CNS) lymphoma
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has known history of, or any evidence of active, non-infectious pneumonitis
* Has evidence of immune- mediated hepatitis, nephritis, or thyroiditis
* Has evidence of interstitial lung disease
* Has evidence of colitis
* Has undergone prior allogeneic hematopoietic stem cell transplantation within the last 5 years
* Requires treatment with a strong CYP3A4 inhibitor/inducer
* Known bleeding disorders
* Requires therapeutic anticoagulation with warfarin or other vitamin K antagonists
* History of stroke or intracranial hemorrhage within 6 months of the first dose of study drug
* Has an active infection requiring intravenous systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is unable to swallow capsules or malabsorption syndrome, disease or condition significantly affecting gastrointestinal function
* Clinically significant cardiovascular disease with uncontrolled arrhythmia, New York Association class 3 or 4 congestive heart failure, history of myocardial infarction within 6 months, or prolonged corrected QT (QTc) > 500 msec
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* Has progressed on prior therapy with ibrutinib or other BTK inhibitors
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days of planned start of study therapy

  * Note: seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2018-11-19 (Actual); Study Completion 2019-01-03 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events assessed using NCI CTCAE version 4 | Up to 5 years
  Summarized based on severity and perceived attribution to study treatment. Will be assessed and tabulated by dose level.
MTD defined as the dose level at which no more than one of 6 patients experiences a dose-limiting toxicity assessed using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4 | Up to 21 days

SECONDARY OUTCOMES:
Complete response rates | Up to 5 years
ORR | Up to 5 years
Overall survival | From study entry to the time of death due to any cause, assessed up to 5 years
  Will be evaluated for each of the cohorts and graphically summarized using the methods of Kaplan and Meier.
Progressive-free survival | From study entry to the time of progression and/or death, assessed up to 5 years
  Will be evaluated for each of the cohorts and graphically summarized using the methods of Kaplan and Meier.

OTHER OUTCOMES:
B, T, and NK cell subtypes | Baseline up to 5 years
  Baseline levels in these markers will be explored in relation to clinical outcome using graphical analyses as well as summarized quantitatively. Will utilize different plotting characters and colors for successes vs. not in the graphical analyses to help identify potential patters, and summarize the changes quantitatively between successes vs not.
Change in biomarker analysis of BTK | Baseline up to 5 years
  Baseline levels in these markers will be explored in relation to clinical outcome using graphical analyses as well as summarized quantitatively. Will utilize different plotting characters and colors for successes versus (vs.) not in the graphical analyses to help identify potential patters, and summarize the changes quantitatively between successes vs not.
Change in biomarker analysis of PD1 | Baseline up to 5 years
  Baseline levels in these markers will be explored in relation to clinical outcome using graphical analyses as well as summarized quantitatively. Will utilize different plotting characters and colors for successes vs. not in the graphical analyses to help identify potential patters, and summarize the changes quantitatively between successes vs not.
Prognostic parameters including ki-67 and cell of origin | Baseline up to 5 years
  Baseline levels in these markers will be explored in relation to clinical outcome using graphical analyses as well as summarized quantitatively. Will utilize different plotting characters and colors for successes vs. not in the graphical analyses to help identify potential patters, and summarize the changes quantitatively between successes vs not.

CONTACTS AND LOCATIONS:
Overall Officials: Kami Maddocks, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu